CLINICAL TRIAL: NCT03153722
Title: Pediatric Ward Discharge Quality Improvement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1016479
Record Dates: First submitted 2017-05-02; First posted 2017-05-15 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Pediatric Hospitalization
Keywords: pediatric; hospital discharge; quality improvement; transition of care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pediatric discharge process intervention (Experimental): All patients hospitalized on the pediatric ward under the pediatric hospitalist service will participate in pediatric discharge process interventions.
  Interventions: Procedure: Pediatric discharge process interventions

INTERVENTIONS:
Procedure: Pediatric discharge process interventions — As this is an iterative quality improvement process, interventions will be evidence-based and chosen to test effectiveness for addressing areas of discharge bottlenecks or inefficiency within our specific hospital's context. Examples of possible interventions may include implementation of a discharge risk assessment (as in Statile et al, Pediatrics 2016), institution of a "medications-in-hand" policy on hospital discharge (as in Sauers-Ford et al, Pediatrics 2016), or initiation of a ward discharge coordinator who will help coordinate outpatient follow-up for patients. Interventions will be implemented in a stepwise fashion, utilizing successive plan-do-study-act cycles, with a minimum 2 month period between interventions to monitor outcomes.

SUMMARY:
This study will utilize an iterative quality improvement process to identify and address delays in the pediatric hospital discharge process.

DETAILED DESCRIPTION:
Hospital crowding has been associated with increased hospital length of stay in pediatric populations and adverse outcomes in adult populations. This study focuses on a 36-bed general pediatric inpatient care unit whose occupancy has seen exponential growth over the past several years. With the growth in patient population, the study hospital is experiencing increasing difficulty with hospital crowding, particularly during key times of year, such as the winter viral respiratory season. During these times, pediatric patients may experience high emergency room wait times, and admitted patients may be required to board in the emergency room or post-anesthesia care unit while they await an inpatient bed. Lack of inpatient bed availability has also, at times, required cancellation of surgical cases and denial of outside hospital patient transfers to the institution, resulting in inconvenience to patients and delays in care.

The pediatric hospital discharge process has come under particular scrutiny as an area in which both the efficiency and the effectiveness of patient care can be improved. Currently, around 10% of patients ready for discharge in a given day from the general pediatric hospitalist service are discharged prior to noon, freeing up this bed space for a new patient. While for some patients, discharge is postponed for medical reasons, others must remain in the hospital for non-medical delays. For example, they may remain hospitalized because they have not yet been seen by a physician, their medications are not available for pick-up from the pharmacy, or they do not have transportation from hospital to home. Several studies in pediatric populations have shown that quality improvement processes can improve discharge efficiency without compromising care quality or patient/family satisfaction. The investigators aim to determine if an iterative quality improvement process can reduce barriers to discharge and therefore decrease pediatric patients' length of stay. They will simultaneously analyze several secondary outcomes to evaluate patient flow, patient/family satisfaction, and subsequent hospital utilization to evaluate for unintended consequences of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Children or young adults less than 21 years of age admitted to the University of California Davis Children's Hospital Pediatric Hospitalist Service on the general pediatric inpatient ward

Exclusion Criteria:

* Adults greater than 21 years of age, including those unable to consent
* Pregnant women
* Prisoners
* Children admitted to other services (i.e. Ear, Nose and Throat Surgery, Pediatric Surgery, Pediatric Gastroenterology, Trauma, Pediatric Nephrology, Pediatric Hematology/Oncology, Pediatric Intensive Care Unit, Neonatal Intensive Care Unit, Newborn Nursery, etc.)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5478 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay index | Time from admission to discharge through study completion in 1 year.
  Length of stay index is a metric that is calculated by Vizient and compares a patient's hospital length of stay to national averages, taking into account the patient's diagnosis, severity of illness, and disease complexity.
Percentage of patients discharged before 1200 | Discharge time for each patient within a 24 hour period on day of discharge.
  Percentage of pediatric hospitalist patients who are discharged before noon on the day they are eligible for discharge.

SECONDARY OUTCOMES:
Readmission | 30 days
  Same hospital 30 day readmission rate
Emergency department re-visit | 7 and 30 days
  Same hospital 7- and 30-day emergency room revisit rate
Patient satisfaction | Mailed to families following hospital discharge through study completion in 1 year.
  Patient/family hospital discharge satisfaction scores, as measured on the Child Hospital Consumer Assessment of Healthcare Providers and Systems (CHCAHPS), which is sent to each family after their child is discharged from the hospital.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lorch SA, Millman AM, Zhang X, Even-Shoshan O, Silber JH. Impact of admission-day crowding on the length of stay of pediatric hospitalizations. Pediatrics. 2008 Apr;121(4):e718-30. doi: 10.1542/peds.2007-1280. PMID 18381501
- [Background] Kostis WJ, Demissie K, Marcella SW, Shao YH, Wilson AC, Moreyra AE; Myocardial Infarction Data Acquisition System (MIDAS 10) Study Group. Weekend versus weekday admission and mortality from myocardial infarction. N Engl J Med. 2007 Mar 15;356(11):1099-109. doi: 10.1056/NEJMoa063355. PMID 17360988
- [Background] Bell CM, Redelmeier DA. Mortality among patients admitted to hospitals on weekends as compared with weekdays. N Engl J Med. 2001 Aug 30;345(9):663-8. doi: 10.1056/NEJMsa003376. PMID 11547721
- [Background] Beck MJ, Gosik K. Redesigning an inpatient pediatric service using Lean to improve throughput efficiency. J Hosp Med. 2015 Apr;10(4):220-7. doi: 10.1002/jhm.2300. Epub 2014 Dec 8. PMID 25483409
- [Background] Statile AM, Schondelmeyer AC, Thomson JE, Brower LH, Davis B, Redel J, Hausfeld J, Tucker K, White DL, White CM. Improving Discharge Efficiency in Medically Complex Pediatric Patients. Pediatrics. 2016 Aug;138(2):e20153832. doi: 10.1542/peds.2015-3832. Epub 2016 Jul 13. PMID 27412640
- [Background] White CM, Statile AM, White DL, Elkeeb D, Tucker K, Herzog D, Warrick SD, Warrick DM, Hausfeld J, Schondelmeyer A, Schoettker PJ, Kiessling P, Farrell M, Kotagal U, Ryckman FC. Using quality improvement to optimise paediatric discharge efficiency. BMJ Qual Saf. 2014 May;23(5):428-36. doi: 10.1136/bmjqs-2013-002556. Epub 2014 Jan 27. PMID 24470173
- [Background] Sauers-Ford HS, Moore JL, Guiot AB, Simpson BE, Clohessy CR, Yost D, Mayhaus DC, Simmons JM, Gosdin CH. Local Pharmacy Partnership to Prevent Pediatric Asthma Reutilization in a Satellite Hospital. Pediatrics. 2016 Apr;137(4):e20150039. doi: 10.1542/peds.2015-0039. Epub 2016 Mar 16. PMID 26983469
- [Derived] Hamline MY, Rutman L, Tancredi DJ, Rosenthal JL; UNIVERSITY OF CALIFORNIA DAVIS CHILDREN'S HOSPITAL DISCHARGE QUALITY IMPROVEMENT WORKING GROUP. An Iterative Quality Improvement Process Improves Pediatric Ward Discharge Efficiency. Hosp Pediatr. 2020 Mar;10(3):214-221. doi: 10.1542/hpeds.2019-0158. Epub 2020 Feb 12. PMID 32051222